CLINICAL TRIAL: NCT03942796
Title: Pregabalin Versus Pulsed Radiofrequency Ablation of Dorsal Root Ganglion for Treatment of Chronic Post Thoracotomy Pain Syndrome
Brief Title: Pregabalin Versus Pulsed Radiofrequency Ablation for Treatment of Chronic Post-thoracotomy Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS/17.12.159
Record Dates: First submitted 2019-05-03; First posted 2019-05-08 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: Chronic Post-thoracotomy Pain
MeSH Terms: interventions — Pregabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lyrica, vronogabic (pregabalin) (Active Comparator): Patients would receive oral pregabalin
  Interventions: Drug: lyrica, vronogabic (pregabalin)
- pulsed radiofrequency ablation of the dorsal root ganglion und (Active Comparator): Patients would receive pulsed radiofrequency ablation of dorsal root ganglion
  Interventions: Procedure: pulsed radiofrequency ablation of the dorsal root ganglion under fluroscopic guidance/ radiofrequency neurolysis/ radiofrequency denervation device name: Neuro Therm TM 1100

INTERVENTIONS:
Drug: lyrica, vronogabic (pregabalin) — Patients would receive oral pregabalin is initiated at a dose of 75 mg twice daily and titrated up to 600 mg as tolerated by the patient at 1,2,3 weeks
  Other Names: lyrica, vronogabic
  Arms: lyrica, vronogabic (pregabalin)
Procedure: pulsed radiofrequency ablation of the dorsal root ganglion under fluroscopic guidance/ radiofrequency neurolysis/ radiofrequency denervation device name: Neuro Therm TM 1100 — Patients would receive pulsed radiofrequency ablation of dorsal root ganglion using the following settings: 2-Hz frequency, 20-ms pulses in a 1 second cycle, 120 second duration and 42°C temperature. Impedance ranges between 150 and 400 Ohms at all levels under fluroscopic guidance. For each pulsed RF application, the procedure will be repeated 4 times, for a total duration of 8 minutes
  Other Names: pulsed radiofrequency ablation of the dorsal root ganglion under fluroscopic guidance/ radiofrequency neurolysis/ radiofrequency denervation
  Arms: pulsed radiofrequency ablation of the dorsal root ganglion und

SUMMARY:
Chronic Post thoracotomy pain syndrome (PTPS) is defined PTPS as pain that develops or increases in intensity after a thoracotomy and persists beyond the healing process, that's to say at least 3 months after the initiating event. The pain has to be localized to the site of incision or, projected to the innervation territory of a nerve situated in this area or referred to a dermatome or Head's zone (after surgery/injury to deep somatic and visceral tissues The incidence of PTPS is 57% and 47% of patients at 3 and 6 months after thoracotomy, respectively.

Management of PTPS begins with prevention. Preventive strategies are based on multimodal preemptive and intraoperative analgesia. Treatment of PTPS is either pharmacologic treatment which is systematically initiated by first line drugs including tricyclic anti-depressants (TCA), serotonin-norepinephrine reuptake inhibitors (SNRI), gabapentinoids. Second-line treatments include topical lidocaine, capsaicin, and weak opioid analgesics (tramadol). Third line treatments consist of strong opioids (oxycodone, morphine) and subcutaneous botilinium toxin injection.

Other therapies for management of CPTP include such modalities as transcutaneous electrical nerve stimulation (TENS), Spinal cord and peripheral nerve stimulation, acupuncture and neurolysis using pulsed radiofrequency for intercostal nerve or dorsal root ganglio and cryoneurolysis for intercostal nerve. The mode of action of pulsed RF is not well-understood, but may include inhibition of excitatory C-fiber responses by repetitive, burst-like stimulation of A-delta fibers, global reduction of evoked synaptic activity and minor structural changes in nerve tissue; elicited by alterations in the function of the blood-nerve barrier, fibroblast activation and collagen deposition.

DETAILED DESCRIPTION:
The aim of the work is to evaluate the effect of oral pregabalin and pulsed radiofrequency ablation (PRF) ablation of the dorsal root ganglion (DRG) in the treatment of chronic post thoracotomy pain syndrome, using Visual Analogue Scale (VAS) score.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status III or IV
* Persistent pain score ≥ 5 on VAS for 3 months or more, not responding to traditional OTC analgesics

Exclusion Criteria:

* Patient refusal
* The presence of pathology that could account for a majority of persistent symptoms (e.g. recurrent cancer)
* coagulopathy
* Uncooperative patients

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Change in the severity of pain | day 1, 3 months
  measured by 11 point VAS score from 0 to 10. the patient is asked to report the severity of his pain in which 0 represents no pain and 10 is the maximum pain. VAS below 5 is considered a "successful" outcome of the treatment method and VAS score ≥ 5 is considered a "failure" outcome. In case of a "failure" outcome, patients will be given oral acetaminophen 500 mg every 8 hours and/or oral ibuprofen 400 mg every 8-12 hours and the need for rescue analgesia will be recorded.
  is measured by 11 point VAS score from 0 to 10. the patient is asked to report the severity of his pain in which 0 represents no pain and 10 is the maximum pain. VAS below 5 is considered a "success" outcome of the treatment method and VAS score ≥ 5 is considered a "failure" outcome. In case of a "failure" outcome, patients will be given oral acetaminophen 500 mg every 8 hours and/or oral ibuprofen 400 mg every 8-12 hours and the need for rescue analgesia will be recorded.

SECONDARY OUTCOMES:
the number of patients who needed rescue analgesia | 2weeks, 1, 2, 3 months
  the Cumulative use of rescue analgesics
the number of patients who developed somnolence as a side effect of treatment | immediately after the intervention, 2weeks, 1, 2, 3 months
  somnolence or excessive daytime sleepiness (EDS) refers to the tendency to fall asleep in inappropriate settings.
the number of patients who developed dizziness as a side effect of treatment | immediately after the intervention, 2weeks, 1, 2, 3 months
  a sensation of unsteadiness accompanied by a feeling of movement within the head
The number of patients who developed nausea as a side effect of treatment | immediately after the intervention, 2weeks, 1, 2, 3 months
  a feeling of sickness with an inclination to vomit.
The number of patients who developed imbalance as a side effect of treatment | immediately after the intervention, 2weeks, 1, 2, 3 months
  the state of being out of equilibrium or out of proportion
The number of patients who developed constipation as a side effect of treatment | immediately after the intervention, 2weeks, 1, 2, 3 months
  a condition in which there is difficulty in emptying the bowels, usually associated with hardened stool.
The number of patients who developed pneumothorax as a side effect of treatment | immediately after the intervention, 2weeks, 1, 2, 3 months
  an abnormal collection of air in the pleural space between the lung and the chest wall, diagnosed by chest xray
Patient satisfaction | 2weeks, 1, 2, 3 months
  Using score including 5-Excellent, 4-Very Good, 3-Good, 2-Fair, and 1-Poor

CONTACTS AND LOCATIONS:
Overall Officials: Gamal M El-Morsy, MD, Study Chair — Professor of Anesthesia and Surgical Intensive Care; Hazem S Maawad, MD, Study Director — Assistant Professor of Anesthesia and Surgical Intensive Care
Locations (1):
- Mansoura University, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting 6 months after publication and for 1 year
Access Criteria: Open access